CLINICAL TRIAL: NCT04002154
Title: Ensayo clínico, Aleatorizado, Abierto, de Grupos Paralelos y Con Grupo Control, Para Explorar la Eficacia Del Gel PAPILOCARE en la reparación de la Mucosa cérvico-vaginal Con Lesiones Causadas Por VPH (Ensayo Clínico PALOMA)
Brief Title: Clinical Trial to Explore the Papilocare Gel Efficacy to Repair the Cervico-vaginal Mucosa With Lesions Caused by HPV
Acronym: PALOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procare Health Iberia S.L. (Industry)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHPC-201501
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Human Papilloma Virus Infection; Human Papilloma Virus; Cervix Lesion
Keywords: HPV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A - papilocare alternative days (Experimental): Arm A: scheme A (21 days / 1 cannula per day + 7 days rest) x 1 month + alternate days up to 6 months (except for menstruation days)
  Interventions: Device: Papilocare vaginal gel
- B - papilocare semiintensive (Experimental): Arm B: scheme B (21 days / 1 cannula per day + 7 days rest) x 3 months + alternate days up to 6 months (except menstruation days)
  Interventions: Device: Papilocare vaginal gel
- C - standard of care (No Intervention): Arm C: usual clinical practice: no treatment

INTERVENTIONS:
Device: Papilocare vaginal gel — Papilocare is a gel vaginally administered by a single-dose cannula. Vaginal gel formulation is effective as a local treatment with controlled systemic absorption and rapid and efficient distribution
  Arms: A - papilocare alternative days; B - papilocare semiintensive

SUMMARY:
Phase II, exploratory, randomized, open, controlled and parallel groups clinical trial to evaluate the effectiveness of exploratory gel Papilocare in the repair of the cervico-vaginal mucosa with lesions caused by HPV. All the patients included in the study will be Randomized (1:1:1).

DETAILED DESCRIPTION:
Phase II, exploratory, randomized, open, controlled and parallel groups clinical trial to evaluate the effectiveness of exploratory gel Papilocare in the repair of the cervico-vaginal mucosa with lesions caused by HPV. All the patients included in the study will be Randomized (1:1:1) to Arm A (Papilocare schedule A), Arm B (Papilocare schedule B) and Arm C (usual clinical practice -without treatment-). Selection period of 1 month, followed by randomization and 6 months of treatment followed by a period of another 6 months without treatment. Patients will visit the site into a total of 5 visits throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Woman between the ages of 30 and 65 (both included).
2. Able to read and understand the Patient Information Sheet and the Informed Consent form.
3. Accept participation in the study and sign the Informed Consent form.
4. Cytological result of ASC-US or LSIL or AG-US, with matching colposcopic image, maximum 3 months before the screening visit.
5. Positive HPV by PCR performed at the screening visit (or positive available at most 3 months prior to the baseline visit).
6. Is capable, at the discretion of the investigator, of complying with the requirements of the study protocol and without impediments to follow the instructions and evaluations throughout it.

Exclusion Criteria:

1. Clinically relevant immune system alterations, or any other autoimmune disease or in treatment with immunosuppressants.
2. Non-diagnosed abnormal genital hemorrhage (during the 6 months prior to the screening visit).
3. To had been vaccinated against HPV.
4. Other symptomatic vulvovaginal infections.
5. Surgical cervical excision in the last year or total hysterectomy.
6. Previous history of gynecological cancer.
7. Participation in any other clinical trial at present or in the 4 weeks prior to the inclusion of the study.
8. Any planned surgery that prevents the correct compliance with the protocol.
9. Use of vaginal contraceptives or other vaginal hormonal treatments.
10. Contraindications for Papilocare gel use or known allergies to any of its components.
11. Women of childbearing age who do not use effective contraceptive methods, pregnant women, with suspicion of pregnancy or woman who are breastfeeding.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Repairment of the cervico-vaginal mucosa in positive HPV women measured by normal cytology with concordant colposcopy image | 6 months
  Evaluate the repairment of the cervico-vaginal mucosa in positive HPV women with a cytological result of squamous atypia of undetermined significance (ASC-US) or low-grade squamous lesion (LSIL) or glandular atypia of undetermined significance (AG-US), with concordant colposcopic image, 6 months after the start of treatment.

SECONDARY OUTCOMES:
Repairment of the cervico-vaginal mucosa in positive HPV women measured by normal cytology with concordant colposcopy image | 3 and 12 months
  Evaluate the repairment of the cervico-vaginal mucosa in positive HPV women with a cytological result of squamous atypia of undetermined significance (ASC-US) or low-grade squamous lesion (LSIL) or glandular atypia of undetermined significance (AG-US), with concordant colposcopic image at 3 and 12 months after the start of treatment.
Reeptielization of the cervico-vaginal mucosa measured by a likert scale. | 3,6 and 12 months
  Evaluate the reeptielization of the cervico-vaginal mucosa months after the start of treatment measured by likert scale, using a total of 5 points (1 is severe ectopy + external bleeding, 2 is severe or extensive ectopy:> 50%, 3 is moderate ectopy: 25-50%, 4 is mild ectopy: <25% and 5 is no ectopy).
Vaginal health status measured by Bachmann Index. | 3,6 and 12 months
  Evaluate vaginal health status from the start of treatment measured by Bachmann Index, it contains 5 domains that evaluate elasticity, type of secretion, pH, epithelial integrity and moisture, scoring each of them from 1 to 5, considering the maximum score as the best vaginal health status.
Satisfaction of papilocare gel use measured by likert scale. | 3 and 6 months
  Evaluate the satisfaction of papilocare gel use by the patients after the start of treatment measured by likert scale, it is a single-item instrument that assesses the degree of satisfaction experienced by the patient with a graded response of 7 values ranging from 1 (satisfied) to 7 (not satisfied at all).
Therapeutic compliance | 3 and 6 months
  Evaluate the therapeutic compliance from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés Bordoy, MD, Study Chair — Hospital os Palma de Mallorca
Locations (9):
- Spain (9):
  - Hospital General Universitario de Alicante, Alicante
  - Clínica Diatros - TEKNON, Barcelona
  - Women´s Health Institute, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Gabinete Médico Velázquez, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Instituto Palacios de Salud y Medicina de la Mujer, Madrid
  - Hospital Quirón Málaga, Málaga

IPD SHARING:
Plan to Share IPD: Yes
It must be discussed with investigators team
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] 2021 ASCCP Poster Presentations. J Low Genit Tract Dis. 2021 Apr 1;25(2S):9-11. doi: 10.1097/LGT.0000000000000602. No abstract available. PMID 33743523